CLINICAL TRIAL: NCT03700905
Title: Multicenter Randomized Controlled Phase III Study of Nivolumab Alone or in Combination With Ipilimumab as Immunotherapy vs Standard Follow-up in Surgical Resectable HNSCC After Adjuvant Therapy
Brief Title: Study of Nivolumab Alone or in Combination With Ipilimumab as Immunotherapy vs Standard Follow-up in Surgical Resectable HNSCC After Adjuvant Therapy
Acronym: IMSTAR-HN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University Hospital, Essen (Other); Westpfalz-Clinical Center GmbH (Unknown); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-934
Record Dates: First submitted 2018-08-03; First posted 2018-10-09 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Intervention Model Description: Arm Ia and Arm Ib are summarized in one Arm, due to central ethics committee, as they both include neoadjuvant and adjuvant treatment compared to Arm II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant/adjuvant Nivolumab and Ipilimumab (Experimental): * Neoadjuvant dose with Nivolumab 3mg/kg after randomization within 2 weeks before surgery
  * Surgical resection of primary tumor including neck dissection according to standard of care
  * 6-7 weeks risk-adapted adjuvant radio(-chemo)therapy 56-66 Gy (chemotherapy Cisplatin 100 mg/m2 on days 1, 22, 43, or Cisplatin once weekly (40mg/m2) for high risk patients only), start within 6 weeks post-surgery
  Arm Ia:
  • Adjuvant administration of Nivolumab 3mg/kg i.v. d1 every 2 weeks within 6 weeks after end of radiotherapy until progression or up to 6 months
  Arm Ib:
  • Adjuvant administration of Nivolumab 3mg/kg i.v. d1 every 2 weeks and Ipilimumab 1mg/kg i.v. d1 every 6 weeks within 6 weeks after end of radiotherapy until progression or up to 6 months
  Interventions: Procedure: Surgical resection of primary tumor; Radiation: Adjuvant radio(-chemo)therapy; Drug: Neoadjuvant Nivolumab; Drug: Adjuvant Nivolumab; Drug: Adjuvant Nivolumab and Ipilimumab
- Surgical resection + adjuvant radio(-chemo)therapy (Active Comparator): * Surgical resection of primary tumor including neck dissection according to standard of care
  * 6-7 weeks risk-adapted adjuvant radio(-chemo)therapy 56-66 Gy (chemotherapy Cisplatin 100 mg/m2 on days 1, 22, 43 or Cisplatin once weekly (40mg/m2) in high risk patients), start within 6 weeks post-surgery
  * Standard follow-up
  Interventions: Procedure: Surgical resection of primary tumor; Radiation: Adjuvant radio(-chemo)therapy

INTERVENTIONS:
Procedure: Surgical resection of primary tumor — Surgical resection of primary tumor including neck dissection according to standard of care
Radiation: Adjuvant radio(-chemo)therapy — Risk-adapted adjuvant radio(-chemo)therapy 56-66 Gy (chemotherapy Cisplatin 100 mg/m2 on days 1, 22, 43, or Cisplatin once weekly (40mg/m2) for high risk patients only)
Drug: Neoadjuvant Nivolumab — Neoadjuvant dose with Nivolumab 3mg/kg after randomization within 2 weeks before surgery
  Arms: Neoadjuvant/adjuvant Nivolumab and Ipilimumab
Drug: Adjuvant Nivolumab — Administration of Nivolumab 3mg/kg i.v. d1 every 2 weeks within 6 weeks after end of radiotherapy until progression or up to 6 months
  Arms: Neoadjuvant/adjuvant Nivolumab and Ipilimumab
Drug: Adjuvant Nivolumab and Ipilimumab — Administration of Nivolumab 3mg/kg i.v. d1 every 2 weeks and Ipilimumab 1mg/kg i.v. d1 every 6 weeks within 6 weeks after end of radiotherapy until progression or up to 6 months
  Arms: Neoadjuvant/adjuvant Nivolumab and Ipilimumab

SUMMARY:
Multicenter randomized controlled phase III study of nivolumab alone or in combination with ipilimumab as immunotherapy vs standard follow-up in surgical resectable HNSCC after adjuvant therapy

DETAILED DESCRIPTION:
Surgically treated locally advanced head and neck squamous cell carcinoma often requires postoperative chemoradiation with high risk of acute and late toxicity. DFS after 2 years is approximately 70%. Combining anti-PD-1 and anti-CTLA4 as a maintenance therapy may improve DFS due to anti-tumor effects of immunotherapy by enhancing cross-presentation of tumor antigens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven SCC of the oropharynx, oral cavity, hypopharynx, and larynx (not older than 3 months before randomization)
* clinical stage III-IVB (T1, N2-3; T2, N2-3; T3, N0-3; T4a, N0-3)
* Oropharyngeal cancer HPV-negative (p16 immunohistochemistry negative)
* Primary tumor and neck metastasis must be resectable
* Written and signed informed consent
* Performance Status of 0 or 1 using ECOG
* Male and female with age ≥ 18
* Curative treatment intent (cM0)
* Screening laboratory values must meet the following criteria and should be obtained within 4 weeks prior to randomization

  * WBC ≥ 2000/μL
  * Neutrophils ≥ 1500/μL
  * Platelets ≥ 100 x103/μL
  * Hemoglobin > 9.0 g/dL
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):
  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
  * AST/ALT ≤ 3 x ULN
  * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Women of childbearing potential (WOCBP)1 must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab.
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product.

Exclusion Criteria:

* Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Patients should be excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
* Prior invasive malignancy except controlled skin cancer or carcinoma in situ of cervix
* Unknown primary (CUP), nasopharyngeal or salivary gland cancer
* Distant metastatic disease or adenopathy below the clavicles
* Serious co-morbidity, e.g. high-grade carotid artery stenosis, congestive heart failure NYHA grade 3 and 4, liver cirrhosis CHILD C. If clinically suspected, further diagnostic is indicated according to the judgement of the investigator.
* Pregnancy or lactation
* Women of child-bearing potential with unclear contraception
* Previous treatment for the study cancer with chemotherapy, radiotherapy, EGFR-targeting agents or surgery exceeding biopsy in head and neck
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to study screening
* Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction: History of severe hypersensitivity reaction to any monoclonal antibody
* History of allergy to study drug components
* Social situations that limit compliance with study requirements or patients with an unstable condition (e.g., psychiatric disorder, a recent history of drug or alcohol abuse, interfering with study compliance, within 6 months prior to screening) or otherwise thought to be unreliable or incapable of complying with the requirements of the protocol
* Patients institutionalized by official means or court order
* Deficient dental preservation status or not accomplished wound healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | approximately 71 months
  disease free survival (DFS) at 3 years of nivolumab alone or in combination with ipilimumab as adjuvant immunotherapy after adjuvant radio(chemo)therapy in locally advanced resected HNSCC

SECONDARY OUTCOMES:
Local regional control (LRC) | Time from randomization to date of first observed histologically proven or death, up to 36 month
  Disease assessment (CT/ MRI) and Panendoscopy and FFPE in case of suspicion or recurrence
Distant metastasis free survival (DMFS) | Time from randomization to date of first observed histologically proven or death, up to 36 month
  Disease assessment (CT/ MRI)
Overall survival (OS) | until end of study (36 months after end of therapy of the last patient), approximately 71 months
  Follow Up- Visits after end of treatment every 3 months until month 36 after randomization, afterwards every 6 months
Acute toxicity and late morbidity | AEs/SAEs should be collected continuously until 12 months after randomization
  Adverse Events Assessment
Quality of life (QoL): QLQ-C30 | through study completion, an average of 3 years
  Questionaire EORTC QLQ-C30
Quality of life (QoL): Questionnaire H&N43 | through study completion, an average of 3 years
  Questionnaire H&N43
Comparison of nivolumab alone group vs control and nivolumab & ipilimumab group vs control in terms of DFS | assessed up to 36 month
  We compare disease free survival, defined as time from randomization to date of first observed either histologically proven recurrence (local, locoregional or distant), or death from any cause whatever occurs first, of arm Ia to arm II and of arm Ib to arm II
Survival depending on PD-L1 Status | after surgery, up to 4 weeks after surgery
  Assessment of PD-L1 Status

CONTACTS AND LOCATIONS:
Overall Officials: PD Dr. med. Chia-Jung Busch, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (7):
- Germany (7):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Technische Universität München, Klinikum rechts der Isar, München, Bavaria
  - Universitätsklinikum Gießen, Giessen, Hesse
  - Klinikum Bielefeld, Bielefeld, North Rhine-Westphalia
  - HELIOS Klinikum Erfurt GmbH, Erfurt, Thuringia
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Katholisches Marienkrankenhaus Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gold KA, Lee HY, Kim ES. Targeted therapies in squamous cell carcinoma of the head and neck. Cancer. 2009 Mar 1;115(5):922-35. doi: 10.1002/cncr.24123. PMID 19156911
- [Result] Cho YA, Yoon HJ, Lee JI, Hong SP, Hong SD. Relationship between the expressions of PD-L1 and tumor-infiltrating lymphocytes in oral squamous cell carcinoma. Oral Oncol. 2011 Dec;47(12):1148-53. doi: 10.1016/j.oraloncology.2011.08.007. Epub 2011 Sep 10. PMID 21911310
- [Result] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Result] Robert C, Long GV, Brady B, Dutriaux C, Maio M, Mortier L, Hassel JC, Rutkowski P, McNeil C, Kalinka-Warzocha E, Savage KJ, Hernberg MM, Lebbe C, Charles J, Mihalcioiu C, Chiarion-Sileni V, Mauch C, Cognetti F, Arance A, Schmidt H, Schadendorf D, Gogas H, Lundgren-Eriksson L, Horak C, Sharkey B, Waxman IM, Atkinson V, Ascierto PA. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2015 Jan 22;372(4):320-30. doi: 10.1056/NEJMoa1412082. Epub 2014 Nov 16. PMID 25399552
- [Result] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank CU, Hamid O, Mateus C, Shapira-Frommer R, Kosh M, Zhou H, Ibrahim N, Ebbinghaus S, Ribas A; KEYNOTE-006 investigators. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32. doi: 10.1056/NEJMoa1503093. Epub 2015 Apr 19. PMID 25891173
- [Result] Seiwert TY, Burtness B, Mehra R, Weiss J, Berger R, Eder JP, Heath K, McClanahan T, Lunceford J, Gause C, Cheng JD, Chow LQ. Safety and clinical activity of pembrolizumab for treatment of recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-012): an open-label, multicentre, phase 1b trial. Lancet Oncol. 2016 Jul;17(7):956-965. doi: 10.1016/S1470-2045(16)30066-3. Epub 2016 May 27. PMID 27247226
- [Result] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Result] Hanna GJ, Adkins DR, Zolkind P, Uppaluri R. Rationale for neoadjuvant immunotherapy in head and neck squamous cell carcinoma. Oral Oncol. 2017 Oct;73:65-69. doi: 10.1016/j.oraloncology.2017.08.008. Epub 2017 Aug 17. PMID 28939078
- [Derived] Zech HB, Moeckelmann N, Boettcher A, Muenscher A, Binder M, Vettorazzi E, Bokemeyer C, Schafhausen P, Betz CS, Busch CJ. Phase III study of nivolumab alone or combined with ipilimumab as immunotherapy versus standard of care in resectable head and neck squamous cell carcinoma. Future Oncol. 2020 Dec;16(36):3035-3043. doi: 10.2217/fon-2020-0595. Epub 2020 Sep 9. PMID 32902312